CLINICAL TRIAL: NCT03595748
Title: Peer Mentorship to Improve Outcomes in Patients on Maintenance Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-8531; R18DK118471 (NIH)
Record Dates: First submitted 2018-06-28; First posted 2018-07-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dialysis
Keywords: Hospitalizations; Dialysis patients; Peer mentorship

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer mentorship intervention (Experimental): This arm of mentees will be assigned to weekly telephone calls with a matched mentor over a period of 3 months.
  Interventions: Behavioral: Peer mentorship
- Usual Care (No Intervention): This arm of mentees will not get a telephone intervention by an assigned mentee

INTERVENTIONS:
Behavioral: Peer mentorship — Participants randomized to this arm of the study will speak with their dialysis peer mentor once a week about fluid intake and adherence to dialysis.
  Arms: Peer mentorship intervention

SUMMARY:
This project tests a peer mentor intervention to improve outcomes in patients with end-stage renal disease (ESRD). The investigators will train peer mentors to deliver social support and to provide information and motivation in order to improve adherence behaviors and self management practices in assigned mentees who are also patients on maintenance hemodialysis. The intervention will consist of a weekly telephone call between mentor and mentee, over a period of 3 months. The study will recruit patients at 7 dialysis facilities (5 in the Bronx, NY and 2 in Nashville, TN) and randomize the patients to the peer mentorship intervention versus usual care. The primary outcome will be the sum of number of emergency department visits and hospitalizations during 3 months of intervention and 9 or 15 months of follow-up observation.

DETAILED DESCRIPTION:
The overarching goal of this research is to improve End Stage Renal Disease (ESRD) related morbidity and mortality. The medical care of patients with ESRD is highly complex and enormously expensive. Hospitalizations drive up to 40% of the cost for ESRD care. Cardiovascular disease and infections account for over 50% of ESRD-related hospitalizations and contribute to disproportionate mortality in this patient population. This study tests the implementation and impact on hospitalization outcomes of a peer mentor led intervention designed to increase effective self-management in patients receiving hemodialysis, in a real-world setting with high potential for widespread dissemination.

Patients receiving hemodialysis who can self-manage their fluid status effectively, are adherent to their dialysis schedule and to their dietary plan are hospitalized less frequently and have lower morbidity and mortality than patients who are less adherent. However, numerous impediments to dialysis self-management exist including facility, physician and patient-level barriers. The following are patient-level barriers to optimal self-management: 1) poor knowledge about the rationale and metrics of estimated dry weight (EDW), 2) poor knowledge about the metrics of urea clearance and nutritional parameters, 3) under-utilization of available hours for unscheduled dialysis, and 4) low self-efficacy leading to non-adherent schedule and dietary behaviors. Dialysis self-management education is often not successful in improving patients' skills. Educational tools from dialysis facilities and providers are didactic, have medical jargon and lack concrete steps to mitigate patient visits to emergency departments (ED) and subsequent hospitalizations. A culturally sensitive, easy to understand educational program that can increase hemodialysis self-management is critically needed.

Peer mentorship has been used effectively to enhance self-efficacy and self-management behaviors in patients with chronic disease. A single study of peer mentorship for ESRD patients found that peer mentors improved adherence and satisfaction with care among mentees. This strategy has high potential to improve the factors that drive hospitalizations among this high-risk patient group. The goal of this research is to implement a peer mentor training program to increase patients' knowledge about the metrics of hemodialysis, enhance self-management to meet EDW, nutritional and adherence goals, and to enhance self-efficacy in mentees. The peer-mentor intervention is based on the information, motivation, behavior (IMB) model of health behavior and the Chronic Disease Self-Management Program. There will be a didactic component to increase knowledge, and a semi-structured component to increase perception of social support. The investigators will test the feasibility of implementation of this program and the efficacy of it to reduce hospitalizations in a pragmatic trial comparing the peer mentor intervention on mentees to a control group assigned to usual care. The study will also test the intervention at two geographically diverse locations (Bronx, NY and Nashville, TN) to provide evidence of its scalability and acceptability in different patient populations. The study hypothesis states: a structured peer mentor telephone intervention will be more effective than usual care in increasing hemodialysis related knowledge, self-management adherent behaviors and in decreasing ED visits and hospitalizations in ESRD.

Specific Aim 1: To evaluate the effects of a 3-month semi-structured and telephone delivered peer mentor intervention on a composite of ED visits and hospitalizations in 100 high risk patients on hemodialysis randomized to peer mentor intervention as compared to 100 high risk patients on hemodialysis assigned to usual care.

* Secondary outcomes include: 1) dialysis adherence (mean weekly minutes of dialysis), 2) mean monthly inter-dialytic weight gain (IDWG), and 3) mean monthly albumin levels, in the intervention mentees as compared to the controls.
* To compare by group patient dialysis knowledge, self-efficacy and social support.

Specific Aim 2: To test the feasibility of a peer training program focused on teaching self-management skills focused on adherence, dietary and fluid management, in dialysis facilities.

* To test the feasibility of a training program conducted in 7 dialysis facilities the investigators will conduct peer training of 20 recruited mentors (10 in New York and 10 in Nashville), using a semi-structured curriculum taught in 4 sets of 2-hour sessions, over 4 weeks per facility.
* To test the fidelity of the curriculum training the investigators will use attendance records, content analysis, pre- and post-knowledge assessments and course evaluations.

This pragmatic trial will test the effects and implementation of a low cost, educational, telephone-based, peer-mentor intervention to increase self-management behaviors of patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years

One of the following:

* One or more hospitalizations or ED visits in the previous month
* >1 missed treatment or 2 shortened dialysis treatments in the last month
* use of catheter as only access
* >4% intradialytic weight gain
* serum albumin less than 3.5 in the last month
* Incident dialysis patient
* Willing to give informed consent and to be randomized and to allow a telephone intervention with mentors
* Speaks Spanish or English

Exclusion Criteria:

* Intellectual disability/ active mental illness or active substance abuse
* less than a 6- month life expectancy
* not a patient at one of the participating dialysis facilities

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine/Montefiore Medical Center, The Bronx, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golestaneh L, Melamed M, Kim RS, St Clair Russell J, Heisler M, Villalba L, Perry T, Cavanaugh KL. Peer mentorship to improve outcomes in patients on hemodialysis (PEER-HD): a randomized controlled trial protocol. BMC Nephrol. 2022 Mar 5;23(1):92. doi: 10.1186/s12882-022-02701-1. PMID 35247960

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Mentors were not included in the trial. Patient participants or mentees were the subjects who were followed for the primary and secondary outcomes. Mentors implemented the intervention.
Period: Overall Study
Arm/Group | Peer Mentorship Intervention | Usual Care
Started | 101 | 98
Completed | 62 | 56
Not Completed | 39 | 42
Not completed — Death | 11 | 12
Not completed — Withdrawal by Subject | 28 | 29
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data available and provided for the 194 participants who completed the protocol.
  Mentors were not included in the trial. Patient participants or mentees were the subjects who were followed for the primary and secondary outcomes. Mentors implemented the intervention.
Groups:
- Peer Mentorship Intervention: This arm of patient participants will be assigned to weekly telephone calls with an assigned mentor over a period of 3 months. They will have observational follow up for 9-15 months thereafter.
  Peer mentorship: Participants randomized to this arm of the study will speak with their dialysis peer mentor once a week about fluid intake, how to improve understanding of and adherence to dialysis.
- Usual Care: This arm of patient participants will not get a telephone intervention by an assigned mentor.
  They will have 12-18 months of observational follow up by study team.
- Total: Total of all reporting groups
Arm/Group | Peer Mentorship Intervention | Usual Care | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.8) | 53.3 (13.8) | 54.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 48 | 46 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 29 | 70
  Not Hispanic or Latino | 51 | 59 | 110
  Unknown or Not Reported | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 59 | 110
  White | 21 | 15 | 36
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 25 | 14 | 39
Region of Enrollment [Number; unit: participants]
  United States | 100 | 94 | 194
Number of hospitalizations in the one year prior to enrollment [Mean (Standard Deviation); unit: Hospitalizations] — Patient self-reported number of hospitalizations in the year prior to enrollment as recorded on baseline assessment.
  Mentors were not included in the trial. Patient participants or mentees were the subjects who were followed for the primary and secondary outcomes. Mentors implemented the intervention
  Hospitalizations | 2.09 (2.66) | 2.27 (2.56) | 2.18 (2.61)
Number of ED visits in the year prior to enrollment. [Mean (Standard Deviation); unit: ED visits] — Patient self-reported number of ED visits in the year prior to enrollment as recorded on baseline assessment.
  Mentors were not included in the trial. Patient participants or mentees were the subjects who were followed for the primary and secondary outcomes. Mentors implemented the intervention
  ED visits | 2.07 (2.75) | 2.11 (2.83) | 2.09 (2.78)

OUTCOME MEASURES:

1. Primary Outcome: ED Visits and Hospitalizations
Description: Each month all enrolled patients will be evaluated for ED visit or hospitalization encounters by both self-report and medical record review. The events will be tabulated each month up to an 18-month period. The rates of the composite event during this period will be determined as event rate per patient-month.
Time Frame: During 3 months of intervention and up to 15 months of follow up (up to 18 months observation total)
Population: Patient participants receiving maintenance dialysis
Measure: Mean (95% Confidence Interval); unit: cases per person-months
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 99 | 95
cases per person-months | 0.244 [0.214 to 0.276] | 0.287 [0.254 to 0.322]

2. Secondary Outcome: Change From Baseline to End of Follow-up in Average Number of Monthly Missed Dialysis Minutes
Description: Average change in number of monthly minutes of dialysis missed by intervention participants as compared to usual care participants over the study period.
Time Frame: up to 18 months
Measure: Mean (Standard Error); unit: minutes per person per month
Groups:
- Intervention Participants: Those participants randomized to receive the intervention, peer mentors calling them weekly for 3 months.
- Usual Care Participants: Those participants randomized to not receiving telephone calls from peer mentors.
Arm/Group | Intervention Participants | Usual Care Participants
Number analyzed (Participants) | 99 | 95
minutes per person per month | 2.4704 (2.146) | 0.3293 (2.122)

3. Secondary Outcome: Change From Baseline to End of Follow-up in Average Monthly Interdialytic Weight Gain in Patient Participants.
Description: Change in monthly average fluid weight gain in-between dialysis treatments by intervention participants as compared to usual care participants over study period.
Time Frame: up to 18 months
Population: Per month rate of increase or decline in mean interdialytic weight gain
Measure: Mean (Standard Error); unit: kg/month
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 99 | 95
kg/month | 0.0061 (0.0464) | -0.0733 (0.0462)

4. Secondary Outcome: Change From Baseline in Average Monthly Serum Albumin Levels
Description: Change in mean monthly albumin levels in intervention mentees as compared to control mentees over follow up period.
Time Frame: up to 18 months
Measure: Mean (Standard Error); unit: g/dL per month
Arm/Group | Intervention Participants | Usual Care Participants
Number analyzed (Participants) | 99 | 95
g/dL per month | 0.0062 (0.0021) | 0.0084 (0.0021)

5. Secondary Outcome: Efficacy of Intervention to Change Dialysis Knowledge in Mentees
Description: Efficacy of intervention to change dialysis knowledge will be assessed based on the Score on Chronic Hemodialysis Knowledge Survey (CHeKs) in patient participants assigned to the peer-mentor intervention as compared patient participants assigned to usual care. Mean change in baseline scores are reported.
  The CHeKs survey consists of 23 multiple choice questions. Total score is determined by summing all correct items (blank items or items with more than one answer are considered incorrect). A positive mean percentage score is indicative of an improvement from baseline and demonstrated increased participant knowledge of hemodialysis care; whereas, a negative mean percentage score is indicative of decrease in demonstrated hemodialysis knowledge.
Time Frame: Baseline and at end of 12-18 months, depending on whether patient enrolled before or after study amendment to shorten follow up time.
Measure: Mean (Standard Error); unit: Percentage Change
Groups:
- Peer Mentorship Intervention: This arm of participants will be assigned to weekly telephone calls with a matched mentor over a period of 3 months.
  Peer mentorship: Participants randomized to this arm of the study will speak with their dialysis peer mentor once a week about fluid intake and adherence to dialysis.
- Usual Care: This arm of participants will not get a telephone intervention by a matched mentor
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
Percentage Change | 0.54 (1.41) | 0.35 (1.5)

6. Secondary Outcome: Efficacy of Intervention to Change Curriculum Specific Dialysis Knowledge in Patient Participants
Description: Efficacy of intervention to change curriculum specific dialysis knowledge in patient participants was assessed based on a change from baseline in score on the "Chronic Hemodialysis Knowledge Survey (CHeKs) Plus" knowledge assessment, an assessment developed by the study team focused on topic covered in mentor training sessions, in patient-participants assigned to intervention as compared patient participants assigned to usual care.
  The CHeKs Plus survey is a multiple-choice training quiz which contains 8 questions. A mean change from baseline score was reported for the groups. A positive mean change demonstrated an improvement in specific hemodialysis knowledge; whereas, a decrease in score is indicative of decrease in specific hemodialysis knowledge.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage Change
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
Percentage Change | 5.21 (2.34) | 1.04 (2.47)

7. Secondary Outcome: Change From Baseline in General Health (GH) Perceptions Domain of V 2.0 of the RAND SF-36 Quality of Life (QOL) in Patient Participants Assigned to Peer-mentor Intervention as Compared to Patient Participants Assigned to Usual Care
Description: Change from baseline in General Health will be assessed using the GH perceptions subscale domain of the RAND SF-36 QoL Health Survey. The GH subscale consists of 5 specific items (Items 1 and 33-36) of the health survey. Item 1 is scored on a 5 point scale ranging from 1 ("Excellent") to 5 ("Very Poor") and items 33-36 are scored on a 5 point scale ranging from 1 ("Definitely True") to 5 ("Definitely False"). Responses are then coded to the RAND scoring key for the respective items as follows: Items 1, 34, and 36 are inversely coded such that a precoded item value of 1 ("Excellent" or "Definitely True") is assigned a final item value of "5" and so forth. Items 33 and 35 maintain the same final item value as precoded item value. This yields an overall scoring range of 5-25 for final value items. No transformation was done. For this measure a mean change from baseline for GH is calculated. A positive mean score is indicative of improved self-perception of general health from baseline.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 2.42 (2.93) | 6.10 (3.24)

8. Secondary Outcome: Change From Baseline in Physical Functioning (PF) Domain of V 2.0 of the RAND SF-36 Quality of Life (QOL) in Patient Participants Assigned to Peer-mentor Intervention as Compared to Patient Participants Assigned to Usual Care
Description: Change from baseline in Physical Functioning (PF) will be assessed using the PF subscale domain of the RAND SF-36 QoL Health Survey. The PF subscale consists of 10 specific items (Items 3-12) of the health survey. These items are scored on a 3 point scale ranging from 1 ("Yes, limited a lot") to 3 ("No, not limited at all") The raw responses values and coded final item values are identical yielding an overall scoring range of 10-30 for final value items. No additional transformation is done. For this measure a mean change from baseline for PF is calculated. A positive mean score is associated with an improved self-perception of physical functioning from baseline.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 0.33 (3.51) | 6.16 (3.90)

9. Secondary Outcome: Change From Baseline in Social Functioning (SF) Domain of V 2.0 of the RAND SF-36 Quality of Life (QOL) in Patient Participants Assigned to Peer-mentor Intervention as Compared to Patient Participants Assigned to Usual Care
Description: Change from baseline in Social Functioning (SF) will be assessed using the SF subscale domain of the RAND SF-36 QoL Health Survey. The SF subscale consists of 2 items (Items 20 and 32) of the health survey. Item 20 is scored on a 5 point scale ranging from 1 ("Not at all") to 5 ("Extremely") and Item 32 is scored on a 5 point scale ranging from 1 ("All of the time") to 5 ("None of the time"). Item 20 is then inversely coded such that a precoded item value of 1 ("Not at all") is assigned a final item value of "5" and a precoded item value of 5 ("Extremely") is assigned a final item value of 1. Item 32 maintains the same final item value as precoded item value. This yields an overall scoring range of 2-10 for final value items. No additional transformation is done. For this measure a mean change from baseline for SF is calculated. A positive mean score is indicative of improved self-perception of physical functioning from baseline.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 1.27 (5.18) | 1.60 (5.71)

10. Secondary Outcome: Effectiveness of Intervention to Change From Baseline to End of Follow-up, Scores on the Perceived Knowledge/Dialysis Self-Management Scale
Description: Effectiveness of intervention to change kidney self-efficacy will be assessed using the "Perceived Kidney/Dialysis Self-Management Scale (PKDSMS)"
  The PKDSMS is a unidimensional eight-item scale used to assess a participant's perceived ability to self-manage their condition. Participant responses are scored on a 1-5 Likert scale, with 1 representing "strongly disagree" to 5 representing "strongly agree." Total scoring ranges from 8-40 with higher scores indicating better perception of self-efficacy and self-management. For this study, mean change from baseline score is reported. A positive mean item score is indicative of better perception of self-efficacy and self-management; whereas, a negative mean item score is indicative of worsening perception of self-efficacy and self-management.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 2.36 (0.77) | 1.01 (1.11)

11. Secondary Outcome: Efficacy of Intervention to Change From Baseline to End of Follow up, Scores on the CESD-R Scale in Participants Assigned to Peer Mentor Intervention as Compared to Participants Assigned to Usual Care
Description: Scores on CESD-R (Center for Epidemiologic Studies Depression Scale Revised) in mentees assigned to intervention as compared to control mentees will be used to assess depressive symptoms.
  CESD. The 20 items in CESD-R scale measure symptoms of depression in nine different groups. The Total CESD-R Score is calculated as a sum of responses to all 20 questions. Response values are as follows:
  Not at all or less than one day = 0 1-2 days = 1 3-4 days = 2 5-7 days = 3 Nearly every day for 2 weeks = 3
  For this study, mean change from baseline score is reported. A positive mean score is indicative of improved depression symptoms; whereas, a negative mean score is indicative of worsening depression symptoms.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | -0.12 (0.07) | 0.05 (0.07)

12. Secondary Outcome: Efficacy of Intervention to Change From Baseline to End of Follow up, Perception of Social Support by Intervention Mentees as Compared to Usual Care Mentees
Description: Perception of social support is measured using scores obtained from the "Multi-dimensional Scale of Perceived Social Support (MSPSS)." The MSPSS is a 12-item scale which measures perceived adequacy of social support from three sources: family, friends, and a significant other. The MSPSS is scored on a 7-point Likert scale (1-7) with 1 representing "very strongly disagree" and 7 representing "very strongly agree" for an overall possible range of 12-84. The total score can also be calculated as a mean score (dividing by 12). Higher scores are indicative of higher perceptions of adequate social support. For this study, change from baseline score of mean score is reported. A positive mean score is indicative of improved perceptions of social support; whereas, a negative mean score is indicative of decreased perceptions of social support.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 0.13 (0.17) | -0.07 (0.18)

13. Secondary Outcome: Efficacy of Intervention to Change From Baseline Kidney Disease Self-management Behaviors in Intervention Mentees as Compared to Usual Care Mentees
Description: Kidney disease self-management was determined by calculating the change in scores from baseline to end of follow up period using the "Kidney Disease Behavioral Index (KDBI)" survey tool. KDBI is a novel 16-item scale based on the Summary of Diabetes Self-Care Activities. It is used measure an individual's self-reported completion of specific self-care activities required for kidney disease self-management.
  The participant is asked to report how often they perform these activities over the past month and the 4-point response options range from 0 = "very slightly or not at all" to 3 = "quite a bit." Scores are summed over the 16 items for a possible scoring range of 0-48, with higher scores indicating a greater engagement in self-care behaviors for kidney disease management. For this study, mean change from baseline score is reported. A positive mean score is indicative of improvement of an individual's completion of specific self-care activities required for kidney disease management.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 1.14 (0.7) | 1.14 (0.7)

14. Secondary Outcome: Efficacy of Intervention to Change From Baseline Kidney Disease Coping Ability in Intervention Mentees as Compared to Usual Care Mentees
Description: The Brief Kidney Cope (Brief "K" [Kidney]-COPE) survey was modified from the Brief COPE for use on study. The Brief K-COPE omits two scales of the full COPE, reduces others to two items per scale, and adds a scale. The Brief K-COPE is intended to foster a wider examination of coping in naturally occurring settings. The Brief K-COPE asks what the participant has done over the past month when a problem taking care of their kidney disease was encountered. The scale consists of 28-items (14 subscales composed of 2 items) scored from 0-3 where "0" = I didn't do this AT ALL, to "3" = I've been doing this A LOT, for a possible scoring range of 0-84. For this study, mean change from baseline score is reported. A positive mean score is indicative of improvement of an individual's ability to cope with their kidney disease; whereas, a negative mean score is indicative a decreased ability to cope with their kidney disease.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | -0.09 (0.09) | 0.86 (0.11)

15. Other Pre Specified Outcome: Efficacy of Intervention to Change From Baseline to End of Follow up, Perception of Dialysis Specific Social Support by Intervention Mentees as Compared to Usual Care Mentees
Description: Change from baseline in Dialysis Specific Social Support was assessed using the Dialysis Specific Support Survey (developed by PI's). This survey was used to characterize the frequency of interactions between the participant and other dialysis patients. This survey consists of 6 items and the total score is the mean of the 6 items. Individual scores for the scale ranged from 1-5 where 1 = ("None of the time") and 5 = ("All of the time"), yielding a possible scoring range of 1-5. For this study, mean change from baseline score is reported. A positive mean score was reflective of more perceived dialysis social support; whereas, a negative mean score was reflective of less perceived dialysis social support.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Peer Mentorship Intervention | Usual Care
Number analyzed (Participants) | 62 | 56
score on a scale | 0.11 (0.12) | 0.17 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment (baseline visit) through 12-18 months of follow up or time at which patient participants and mentees were censored.
Description: Participants with hospitalizations or ED visits. Non-serious adverse events were only collected for those instances where:
  1. There was embarrassment and/or stigma related to being identified as a high-risk patient
  2. Distress related to concern for loss of privacy of health information by mentor disclosure
  3. Distress related to telephone conversations with mentors
  The trial examined outcomes in patient participants and not mentors. Mentors implemented the intervention: peer mentorship.
Arm/Group | Peer Mentorship Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 11/99 | 15/95
Serious Adverse Events (participants affected / at risk) | 64/99 | 66/95
Other Adverse Events (participants affected / at risk) | 0/99 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Mentorship Intervention (N=99) | Usual Care (N=95)
Hospitalization (Surgical and medical procedures) | 64 (171) | 66 (194)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03595748/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03595748/ICF_001.pdf